CLINICAL TRIAL: NCT00177541
Title: Further Enhancing Non-pharmacologic Therapy for Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Neil Resnick, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5R01AG020629-02 (NIH); 5R01AG020629-02 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Urge Urinary Incontinence
Keywords: urge incontinence; biofeedback; pelvic floor muscle training; behavior modification
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biofeedback (Experimental): Biofeedback assisted pelvic floor muscle therapy (3 visits)
  Interventions: Behavioral: Biofeedback, pelvic floor muscle training, fMRI

INTERVENTIONS:
Behavioral: Biofeedback, pelvic floor muscle training, fMRI — Biofeedback, pelvic floor muscle training, fMRI

SUMMARY:
To determine the mechanisms mediating the therapeutic efficacy of pelvic floor muscle exercises and biofeedback for urge urinary incontinence, as well as the characteristics of patients most likely to respond. By identifying the key components of this treatment, we hope to simplify it and make it more easily applicable, more effective, less expensive, and thus more useful for people with urge incontinence in the future.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is prevalent and morbid in the elderly, and its associated costs exceed $26 billion annually. Although effective therapy exists, it is underutilized. This is particularly true for non-pharmacologic therapies, which are at least as effective as drugs but safer, and recommended as the initial approach by every national panel. If therapies such as biofeedback (which targets pelvic muscles and detrusor suppression) are to become more widely used, they will require simplification, fewer and briefer sessions, less expensive equipment, and less sophisticated therapists. Unfortunately, such protocols cannot yet be devised because it is unknown which components are essential. We postulate that the mechanisms mediating effectiveness can be identified and that such knowledge will make it possible to enhance efficacy and to formulate more feasible and cost-effective protocols. Since reduction in UI correlates weakly with improved quality of life, however, it is important that biofeedback's impact on life quality be assessed concomitantly to ensure that formulation of such streamlined methods does not eliminate components essential for improved quality of life, even if they have no physiological correlates. We will address these issues by treating at least 150 elderly subjects with urge UI in an 8-week course of biofeedback. We will collect clinical and quality of life data and perform extensive physiologic testing on each subject at baseline and 8 weeks later. Improvement will be correlated with change in physiologic and quality of life parameters to identify the parameters that likely mediated it. Knowledge from this study should identify predictors and mechanisms mediating success of biofeedback; suggest ways that it could be further improved; facilitate development of less expensive, quicker, and more feasible protocols to deliver it (potentially permitting application to less motivated or cognitively impaired patients); and shed insight into mechanisms that may even improve efficacy of other interventions.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory women over age 60, who are incontinent at least twice weekly for 3 months despite correction of potentially reversible causes.
* urinary incontinence (urge or predominantly urge) by clinical criteria.
* able to accurately complete a voiding diary, to perform a 24-hour pad test under direction, and to undergo instruction in biofeedback.

Exclusion Criteria:

* significant mental impairment [mini mental status exam (MMSE) ≤ 20)
* urethral obstruction
* history of bladder cancer
* spinal cord lesions
* multiple sclerosis
* pelvic radiation
* interstitial cystitis
* artificial sphincter implant
* expected to have changes in medications/doses during the trial
* medically unstable
* Patients with factors that could cause transient UI [e.g., current urinary tract infection (UTI), acute confusion] will be treated in concert with the subject's primary care provider and considered for enrollment if their UI persists.
* conditions that require endocarditis prophylaxis (such as heart valve problems or bacterial endocarditis)
* being unable to undergo fMRI because of claustrophobia or any metallic objects in the body, such pacemakers, metallic prostheses, aneurism clips or others.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2004-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Percentage reduction in urge incontinence episodes at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Various urodynamic parameters such as, e.g.: | 12 weeks
Increase in functional bladder capacity at 12 weeks | 12 weeks
Volume at first detrusor overactivity at 12 weeks | 12 weeks
Improvement in QoL at 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil M Resnick, MD, Principal Investigator — University of Pittsburgh; Becky Clarkson, PhD, Study Director — University of Pittsburgh
Locations (1):
- Geriatric Continence Research Unit, NE547 Montefiore UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Burgio KL, Locher JL, Goode PS, Hardin JM, McDowell BJ, Dombrowski M, Candib D. Behavioral vs drug treatment for urge urinary incontinence in older women: a randomized controlled trial. JAMA. 1998 Dec 16;280(23):1995-2000. doi: 10.1001/jama.280.23.1995. PMID 9863850
- [Background] Resnick NM. Improving treatment of urinary incontinence. JAMA. 1998 Dec 16;280(23):2034-5. doi: 10.1001/jama.280.23.2034. No abstract available. PMID 9863856
- [Derived] Resnick NM, Perera S, Tadic S, Organist L, Riley MA, Schaefer W, Griffiths D. What predicts and what mediates the response of urge urinary incontinence to biofeedback? Neurourol Urodyn. 2013 Jun;32(5):408-15. doi: 10.1002/nau.22347. Epub 2012 Nov 20. PMID 23168606